CLINICAL TRIAL: NCT03909815
Title: Do Dual Mobility Cups Prevent Dislocation After Total Hip Arthroplasty Performed Due to Femoral Neck Fracture? A Registry-based, Pragmatic, Randomized Controlled Trial Comparing Dual Mobility With Standard Cups
Brief Title: Dual Mobility Cups in Hip Fracture Patients
Acronym: DUALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-101; ISRCTN11895196 (Registry Identifier: The UK's Clinical Study Registry)
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Femoral Neck Fractures
Keywords: total hip arthroplasty; dual mobility cup; dislocation; mortality; periprosthetic joint infection; health economy
MeSH Terms: conditions — Femoral Neck Fractures; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Insertion of dual mobility cup
  Interventions: Device: Dual mobility cup
- Control (Active Comparator): Insertion of standard cup
  Interventions: Device: Standard cup

INTERVENTIONS:
Device: Dual mobility cup — Patients with a displaced femoral neck fracture eligible for THA receive a dual mobility cup, as opposed to a standard cup in the control group.
  Arms: Intervention
Device: Standard cup — Patients with a displaced femoral neck fracture eligible for THA receive a standard cup, as opposed to a dual mobility cup in the experimental group.
  Arms: Control

SUMMARY:
Our aim is to develop a strategy that reduces the risk of dislocations after total hip arthroplasty surgery performed due to femoral neck fracture. We therefore perform a register-nested, pragmatic, randomized controlled trial to investigate the safety and efficacy of dual mobility cups that were designed to minimize the risk of dislocation in the large and fragile group of elderly patients with femoral neck fractures.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is regularly performed in patients with a femoral neck fracture. However, dislocation is very common after THA in hip fracture patients, and this complication is deleterious to health and quality of life. The dual mobility cup offers a technical solution that potentially reduces the risk of dislocation. There is however no high-level evidence to support the general use of dual mobility cups in patients with displaced femoral neck fractures, and the purpose of the proposed study is to provide evidence to support or refute the use of this concept in the very large group of hip fracture patients.

We a register-nested, pragmatic randomized controlled trial (RCT) to investigate the safety and efficacy of dual mobility cups that were designed to minimize the risk of dislocation after THA. Our aim is thus to investigate whether the incidence of dislocations after THA surgery performed due to femoral neck fracture can be reduced by the use of this device.

The intervention group receives a dual mobility cup (of any brand that is in general use in Sweden), and the control group receives a standard cup (of any brand that is in general use in Sweden). The choice of cup or stem fixation (cemented or uncemented), femoral head size, brand of stem type, surgical approach, antibiotic prophylaxis, and postoperative mobilization are up to the surgeon's choice and the routines that are relevant at each study site.

The necessary infrastructure for this register-nested RCT is present within the Swedish Hip Arthroplasty Register (SHAR) and the Swedish Fracture Register (SFR). Pre-operative registration of fractures is already established within the SFR, and an online platform to screen, include and randomize eligible patients is established. Cross-matching of data from the SFR and the SHAR with the database of the Swedish Patient Register (SPR) is performed in order to catch endpoint not routinely collected by the SHAR.

Expanded recruitment in collaboration with UK, WHITE 12-Duality, started 10/09/2022. https://www.isrctn.com/ISRCTN11895196

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis: displaced femoral neck fracture type AO 31-B2 or B3/Garden type 3 or 4
* Eligible for THA according to local guidelines and routines

Exclusion Criteria:

* Previous inclusion of contralateral hip
* Delayed fracture surgery (date of injury >7 days prior to date of randomization)
* Pathological or stress fracture of the femoral neck, or fracture adjacent to a previous ipsilateral hip implant
* Inability or unwillingness to give written consent
* Dementia (as diagnosed by the screening physician)
* Unavailability of both interventions for a study subject (e.g., implants being out of stock, or lack of the individual surgeon's expertise to perform either procedure)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Dislocation | 1 year after index surgery
  Dislocation will be ascertained by identifying the occurrence of any closed or open reduction of the previously inserted THA (the "index joint") within one year after surgery.

SECONDARY OUTCOMES:
Any re-operation of the index THA | 1 year after index surgery
  Re-operation will be defined as the occurrence of any surgical procedure performed on the previously treated hip within one year after surgery.
Periprosthetic joint infection | 1 year after index surgery
  Periprosthetic joint infection will be defined as the occurrence of any sign of deep infection around the previously inserted THA within one year after surgery, defined by registration of ICD or NOMESCO codes.
Patient-reported outcome | 1 year after index surgery
  Patient-reported outcome as assessed by EQ-5D-VAS (routinely collected by the SFR at index surgery in order to obtain pre-trauma baseline, and 1 year post-operatively)
Short-term mortality | 90 days after index surgery
  90-day mortality, as registered in the NPR
Medium-term mortality | 365 days after index surgery
  365-day mortality, as registered in the NPR
Cost-effectiveness | 1 year after index surgery
  Procedural costs for intervention and control treatment will be recorded at all sites, ensuring documentation of baseline costs for the two treatment alternatives. Procedural costs of admissions for closed reductions as well as for reoperations will also be collected from all units.

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Lazarinis, MD, PhD, Study Chair — Uppsala University Hospital
Locations (2):
- Nils Hailer, Uppsala, Sweden
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolf O, Mukka S, Notini M, Moller M, Hailer NP; DUALITY GROUP. Study protocol: The DUALITY trial-a register-based, randomized controlled trial to investigate dual mobility cups in hip fracture patients. Acta Orthop. 2020 Oct;91(5):506-513. doi: 10.1080/17453674.2020.1780059. Epub 2020 Jun 22. PMID 32567472